CLINICAL TRIAL: NCT07376668
Title: WhatsApp-assisted Prehabilitation Programme for Adult Patient Undergoing Elective Colorectal Cancer Surgery - A Randomised Controlled Trial
Brief Title: Effects of a WhatsApp-assisted Prehabilitation for Patient Undergoing Elective Colorectal Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tseung Kwan O Hospital, Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, SUNG HOI LING SHERING, Principal Investigator, Tseung Kwan O Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIRB-2025-099-2
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer (Diagnosis)
Keywords: Prehabilitation
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — Methods; Preoperative Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: A computer-based randomization will be utilized to allocate patients into either one group. Eligible participants will be randomly assigned in a 1:1 ratio to either control group or intervention group. Block randomization was performed through a computer-generated sequence, and serial and opaque with sealed envelopes will be prepared in by independent staff not involved in clinical care or screening or assessment, in which will be used to conceal the sequence until the intervention as assigned at the outpatient preoperative clinic. A single blinded with outcome assessor will be conducted in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp-assisted prehabilitation (Experimental): Patient will receive WhatsApp-assisted prehabilitation plus standard care
  Interventions: Other: Intervention; Other: Standard care
- Standard care (No Intervention)

INTERVENTIONS:
Other: Intervention — In addition to standard care, participants will receive digital approach of WhatsApp-assisted prehabilitation programme and then start the home-based training for about 3-4 weeks prior to the surgery. The WhatsApp-assisted prehabilitation includes exercises training, dietary advice and psychological support. Contents will contain elements of physical training (e.g. aerobic and resistance exercises) and psychological therapy (e.g. meditation) will be delivered through WhatsApp at three sessions (day 1, 3 & 5) per week for 30 minutes and 15 minutes respectively, educational information associated with colorectal cancer surgery and prehabilitation(e.g. high risks factors towards surgical complications) and dietary advices (e.g. recipes) will be delivered on weekly
  Other Names: Prehabilitation
  Arms: WhatsApp-assisted prehabilitation
Other: Standard care — Standard care as per department guidelines with ERAS protocol (including smoking cessation program, preoperative counselling, early rehabilitation program)
  Arms: WhatsApp-assisted prehabilitation

SUMMARY:
The goals of this study is to evaluate the feasibility and the effects of a WhatsApp-assisted prehabilitation for colorectal cancer patients undergoing elective surgery. The main questions are: If the digital prehabilitation is feasible and acceptable by the colorectal cancer patient prior to elective surgery? If this prehabilitation helps to improve the postoperative complications, length of stay, physical activity and psychological well-being for colorectal cancer patients receiving surgery.

Researcher will compare the prehabilitation plus standard care to standard care only to see if the prehabiliation helps the colorectal cancer patients.

Participants will: 1) enrolled in a approximate 4 weeks (3 episodes/ week) prehabilitation program containing educational information of colorectal cancer, dietary advice, exercises training and psychological podcasting. 2) will answer the survey weekly and after surgery. 3) keep the standard care as per department guidelines

DETAILED DESCRIPTION:
Colorectal cancer ranks the second most prevalent forms of cancer in Hong Kong and surgery is still the primary curative option. Although compromising result of shorten general length of stay (LOS) in enhanced recovery after surgery (ERAS) protocol is illustrated, surgical complications such as postoperative ileus (POI) remain unresolved and significant burden associated leads to suboptimal patients' outcomes of prolonged LOS and physical deconditioning with extended rehabilitation. Prehabilitation refers to optimization in a single or multi-disciplinary approach of exercises training, nutritional therapy and psychological counselling, improves physical fitness, strengthens cardiopulmonary function and reduce mental distress through lifestyle modification and better physiological reserve. However, the concept of educations in form of preoperative exercises and nutritional counselling outweighs the purposes of actual prehabilitation and short-handed allied health professionals limited accessibility of regular out-patient counselling in the current clinical practices. Consequently, poor adherence to these preoperative trainings may result in to poor surgical outcomes.

A single with assessor-blinded, double-armed randomised controlled trial study with a prior pilot will be employed to examine the feasibility and effects of a technology-assisted prehabilitation for patients with colorectal cancer surgery. Outcomes of postoperative complications, LOS, physical activity, nutritional status, gastrointestinal recovery and psychological well-being will be evaluated. Elective colorectal cancer surgery patient will be invited to participated in this study.

The result will provide insights of the use of digital approach. To our knowledge, this is the very first trial of digital prehabilitation for CRC patients in Hong Kong public hospitals. Therefore, it provides positive contribution and acts as an important quality benchmark for patients' outcomes. The findings will also generate knowledge on the optimalization of care provided to CRC patients prior to surgery and assist to develop a structured and effective health system in our community. This innovation may have implications to other research studies and extends the potential clinical practices to related subspecialities such as gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of colorectal-related cancer
* scheduled for elective colorectal cancer surgery as primary treatment
* aged 18 years or above
* expected surgery date more than 21 days
* able to collaborate in the study and sign the informed consent
* able to use WhatsApp application

Exclusion Criteria:

* identified or known premorbid, that inability to follow the programme
* able to understand written and spoken Cantonese/ Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Postoperative period: assessed up to first year postoperative
  measured by the Comprehensive Complication Index (CCI), which integrates in a single formula all complications by severity, ranging from 0 (uneventful course) to 100 (death).

SECONDARY OUTCOMES:
Length of hospital stay (LOS) | Postoperative period: assessed up to the first year postoperative
  to evaluate the length of postoperative hospital stay
Physical activity | Assessments at baseline, weekly before the surgery and on the day of discharge: assess up to first year postoperative
  measured by the International Physical Activity Questionnaire Short Form (IPAQ-SF), seven items were assessed in frequency and duration over the past seven days, categorizing it into four types: vigorous intensity, moderate intensity, walking, and sitting. An average metabolic equivalents score (MET, min·w-1) was calculated to assess total physical activity as well as for each type of activity, separately. For walking activities, all types of walking were included and an average MET score was derived. The same procedure was carried out for medium intensity and high intensity activities. By calculating the number of activity days multiplied by the average duration per activity, statements about the energy consumption per week and the fitness level can be derived.
Gastrointestinal recovery | Postoperative period: assessed up to 30 days postoperative
  measured as time to first flatus (in hours)
Gastrointestinal function | Postoperative period: assess up to 30 days postoperative
  measured as time to first bowel (hours)
Anxiety and depression | Assessments at baseline and on the day of discharge: assess up to first year postoperative
  assessed by the Chinese version of Hospital Anxiety and Depression Scale (C-HADS), a 14-question measure with seven items each for depression and anxiety. HADS generates separate scores for anxiety and depression as well as a combined score of psychological distress. Continuos variable 0-21 (0-7 normal value, 11-21 anxiety/depression), higher value from baseline will represent a worse outcome.
Quality of health-related life | Assessments at baseline and on the day of discharge: assess up to first year postoperative
  evaluated by the Short Form 12 Health Survey (SF-12 version 2 (Hong Kong)), with Physical Component Summary (PCS) and Mental Component Summary (MCS). Scores range from 0-100 for the 8 underlying health domains, with higher scores meaning better Health-Related Quality of Life (HRQoL)

OTHER OUTCOMES:
Adherence to the prehabilitation | From enrollment to the completion of study up to 18 months
  percentage of completed at least 75% of the prehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: SHERING SUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Tseung Kwan O Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07376668/Prot_SAP_000.pdf